CLINICAL TRIAL: NCT00547001
Title: A Comparison of Hormonal Therapy: Tapering Regimens for Mediating Hot Flashes
Brief Title: Comparison of Hormonal Therapy: Mediating Hot Flashes Tapering Regimens for Mediating Hot Flashes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Peter Schnatz, MD - Principal Investigator, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCHN002140HI
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Hot Flashes; Night Sweats
Keywords: Menopause; Hot flashes; vasomotor symptoms; tapering regimen; hormonal therapy; Other menopausal symptoms including mood changes
MeSH Terms: conditions — Hot Flashes | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Group A will be tapered over 4 weeks, starting at baseline (week 0). Subjects in this group will take one tablet of ET daily (effective dose, 0.75 mg) for week 1, then one 0.50 mg tablet daily for week 2, then one 0.25 mg tablet daily for week 3, and finally one 0.125 mg tablet daily for week 4.
  Interventions: Drug: Estradiol
- 2 (Placebo Comparator): Group B will be administered placebo. These tablets will appear identical to those administered to subjects in Group A, but the tablets will contain no estrogen. Subjects in this group will be instructed to take one pill every day for the 4 weeks. Thus, while patients will, in effect, be stopped abruptly from their therapy, there is still the potential of a placebo effect.
  Interventions: Drug: Estradiol
- 3 (No Intervention): Group C will have their therapy discontinued acutely at baseline (week 0); i.e., these subjects will not take any tablets after the 8-week stabilization phase ends. While we recognize that this group will not be blinded to the regimen they are receiving, we feel that group C will be important to include in light of the consistent decrease in vasomotor symptoms experienced by women taking placebo. Because women taking placebo have approximately a 35% decrease in vasomotor symptoms, it will be important to compare our taper regimen to the "real life" scenario of stopping medication abruptly.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — 1mg during stabilization & then a taper to 0.75mg, 0.5mg, 0.25mg, 0.125mg.

SUMMARY:
This study will evaluate whether there is a difference in the proportion of women who report a worsening severity of their hot flashes between three tapering schedules for one accepted HT/ET regimen. Secondarily, we hope to evaluate whether there is a difference in the frequency (number of occurrences per week), severity (defined as a subjective scale mild, moderate, or severe), and "Severity Index" (SI, equaling the product of both) of hot flashes between three tapering schedules for one accepted HT/ET regimen.

DETAILED DESCRIPTION:
A Comparison of Hormonal Therapy:

Tapering Regimens for Mediating Hot Flashes

Clinicians have been asking for years whether a tapering dose of HT would make a difference in the frequency and severity of vasomotor symptoms after menopausal women stop HT therapy. This planned randomized, placebo-controlled trial (RCT) seeks to evaluate whether there is a difference in the proportion of women who report a worsening severity of their hot flashes between three tapering schedules for one accepted HT/ET regimen. Secondarily, we hope to evaluate whether there is a difference in the frequency (number of occurrences per week), severity (defined as a subjective scale mild, moderate, or severe), and "Severity Index" (SI, equaling the product of both) of hot flashes between three tapering schedules for one accepted HT/ET regimen.

All participants will be randomized to one of the three arms (taper arm, placebo arm, and "cold turkey" arm). Each patient's gynecologist will be aware of the patient's involvement in the study and will assist by providing baseline safety information. All patients will be taken off their current HT/ET regimen and will be placed on study medication (1 mg of Estradiol PO every day for 8 weeks, "stabilization" phase). After the 8-week stabilization period, all participants will begin the therapy corresponding to the arm to which they were randomized. Each patient in the taper or placebo arm will take one capsule per day. The patients in the "cold turkey" arm will discontinued acutely after the stabilization.

The patients will keep a diary of the number and frequency of symptoms during the study. Patients will be contacted by phone to confirm that they are completing their diaries and that they have not developed side effects or complications that could force their discontinuation from the study.

Patients will be followed for several additional weeks, after discontinuation from treatment or placebo, to monitor for symptoms. At the end of the study, our coordinator will contact the patient to assure that Medroxyprogesterone acetate, MPA, was taken properly by those women who have a uterus. They will also confirm that no other symptoms, complications, or questions have arisen. At that time, they will be able to return to their prior therapy as deemed appropriate by them and their physician.

Patients will be recruited by invitation upon presenting for care to their physician. With invitations at recruitment, all patients will be given a study form. Reasons for ineligibility or refusal will be noted. After expressing interest, the physician or practice of record will sign a form acknowledging that their patient has had an annual physical exam (including pelvic exam) within the last 12 months and that a mammogram has been reported as negative (BIRADS I or II) within the last 24 months. An appointment will be made with one of our study personnel or coordinators. The patient will bring the signed form to this visit. At this enrollment / consent visit, their eligibility criteria will be reviewed. All patients will sign the informed consent, and be randomized to a group.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* ages 35-70, inclusive.
* Postmenopausal (Natural or surgical: see definitions).
* Currently on HT/ET for at least 6 months for vasomotor symptomatology.
* Vasomotor symptoms are currently controlled on medication .
* An annual physical & pelvic exam has been performed within the last 12mo
* The patient has had a normal mammogram(BIRADS I/II) within the last 24mo

Exclusion Criteria:

* Males
* Hypertension, defined as either SBP >140 mmHg or DBP >90 mmHg
* Lack of compliance (willingness to adhere to protocol)
* Inability or unwillingness to swallow pills
* Patients with any contraindications to HT/ET

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2007-08; Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether there is a difference in the proportion of women who report a worsening severity of their hot flashes between three tapering schedules for one accepted HT/ET regimen. | During the tapering and post taper time period.

SECONDARY OUTCOMES:
frequency, severity, and "Severity Index" of hot flashes. | During the tapering and post taper time period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter F. Schnatz, D.O., Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States